CLINICAL TRIAL: NCT00756119
Title: Measurement of Cardiac Output and Blood Volumes Using Transonic Ultrasound Dilution Technology - Clinical Evaluation and Validation
Brief Title: Measurement of Cardiac Output and Blood Volumes Using Transonic Ultrasound Dilution Technology
Status: Completed | Type: Observational
Sponsor: Transonic Systems Inc. (Industry)
Collaborators: Russian Academy of Medical Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: TSI-R-COstatus-1A-H
Record Dates: First submitted 2008-09-17; First posted 2008-09-19 (Estimated); Last update posted 2012-05-31 (Estimated); Status verified 2012-05

CONDITIONS: Post Cardiac Surgery Patients

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Measurement of the amount of blood pumped by the heart (cardiac output) and blood volumes in sick patients is important for doctors to better treat these patients. Current procedures available demand difficult invasive procedures and hence these parameters are not measured with enough frequency and are also limited to certain patients. The new COstatus system is capable of using the already existing arterial and venous lines placed in critically ill patients and thus provides an opportunity to measure these parameters less invasively and with enough frequency.

The purpose of this study is to measure cardiac output and blood volumes using ultrasound dilution technology (COstatus system)in post cardiac surgery adult patients and compare the cardiac output measurements with a current clinical reference method, thermodilution.

ELIGIBILITY:
Inclusion Criteria:

* Post cardiac surgery adult patients
* Patients with heart catheter and arterial catheter

Exclusion Criteria:

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Post cardiac surgery adult patients
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2006-12; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alexsandr A Eremenko, MD, Principal Investigator — Russian Academy of Medical Sciences
Locations (1):
- National Research Center of Surgery, Russian Academy of Medical Sciences, Moscow, Moscow, Russia

REFERENCES:
- [Background] Eremenko A, Balykov I, Chaus N, Kislukhin V, Krivitski N. Use of an extracorporeal arteriovenous tubing loop to measure cardiac output in intensive care unit patients by ultrasound velocity dilution. ASAIO J. 1998 Sep-Oct;44(5):M462-4. doi: 10.1097/00002480-199809000-00028. PMID 9804473
- [Background] Eremenko AA, Chaus NI, Kislukhin VV, Balykov IV. [The determination of cardiac output by the dilution of ultrasonic blood density]. Anesteziol Reanimatol. 1998 Jul-Aug;(4):4-6. Russian. PMID 9770808
- [Background] Krivitski NM, Kislukhin VV, Thuramalla NV. Theory and in vitro validation of a new extracorporeal arteriovenous loop approach for hemodynamic assessment in pediatric and neonatal intensive care unit patients. Pediatr Crit Care Med. 2008 Jul;9(4):423-8. doi: 10.1097/01.PCC.0b013e31816c71bc. PMID 18496416